CLINICAL TRIAL: NCT00571675
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter, Phase 2 Study Comparing AT-101 in Combination With Docetaxel and Prednisone Versus Docetaxel and Prednisone in Men With Chemotherapy-Naïve Metastatic Hormone Refractory Prostate Cancer (HRPC)
Brief Title: A Study Comparing AT-101 in Combination With Docetaxel and Prednisone Versus Docetaxel and Prednisone in Men With Chemotherapy-Naïve Metastatic Hormone Refractory Prostate Cancer (HRPC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ascenta Therapeutics (Industry)
Responsible Party: Melissa Brookes, Sr. Project Manager, Clinical Development, Ascenta Therapeutics
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AT-101-CS-205
Record Dates: First submitted 2007-12-11; First posted 2007-12-12 (Estimated); Last update posted 2010-11-09 (Estimated); Status verified 2010-11

CONDITIONS: Hormone Refractory Prostate Cancer
Keywords: Prostate Cancer; Hormone Refractory Prostate Cancer; HRPC; Docetaxel; Taxotere; Prednisone; Metastatic (Stage IV) Disease; Chemotherapy-naïve metastatic Hormone Refractory Prostate Cancer (HRPC)
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm Metastasis; Disease | interventions — gossypol acetic acid; Prednisone; Docetaxel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): AT-101, prednisone and docetaxel
  Interventions: Drug: AT-101, prednisone and docetaxel
- 2 (Placebo Comparator): Placebo, prednisone and docetaxel
  Interventions: Drug: placebo, prednisone and docetaxel

INTERVENTIONS:
Drug: AT-101, prednisone and docetaxel — docetaxel (75mg/m2 intravenously over 1 hour on day 1, every 21 days [one cycle]), oral prednisone (5mg BID on days 1-21), and oral AT-101 on cycle days 1-3
  Arms: 1
Drug: placebo, prednisone and docetaxel — docetaxel (75mg/m2 intravenously over 1 hour every 21 days [one cycle]), oral prednisone (5mg BID on days 1-21), and oral placebo on cycle days 1-3
  Arms: 2

SUMMARY:
This is a randomized, double-blind, placebo-controlled, multinational Phase 2 study to evaluate and compare oral AT-101 in combination with docetaxel and prednisone versus docetaxel and prednisone plus placebo in the treatment of chemotherapy-naïve metastatic hormone-refractory prostate cancer, who have received hormonal therapy but not chemotherapy.

DETAILED DESCRIPTION:
Further Study Details provided by Ascenta.

ELIGIBILITY:
Inclusion Criteria:

1. Males age ≥ 18 years with histologically confirmed adenocarcinoma of the prostate, which is now metastatic (e.g. any T, any N, M1a-c) based on bone scan, CT scan, or MRI scan.
2. Progression of disease despite androgen deprivation (androgen ablation or surgical castration) and anti-androgen withdrawal as documented by one or more of the following.

   * Progression of measurable disease per RECIST
   * Bone scan progression, defined as the appearance of ≥ 2 new lesions on bone scan, attributable to prostate cancer
   * Rising PSA, as defined by increasing levels on at least two consecutive assessments, following a prior assessment taken as a reference value, where all of the following are met:

     * The assessments are at least one week apart, with the first assessment at least one week later than the reference value
     * Progressive increase in the two assessments after the reference value, without an intervening decrease between assessments.
     * The last value prior to study entry is ≥ 2 ng/mL
3. Serum testosterone level ≤ 50 ng/dL post orchiectomy or while maintained on continuous or intermittent medical androgen suppression with a LHRH agonist or antagonist.
4. At least 2 weeks since ketoconazole or systemic steroids (any dose); 2 weeks since prior flutamide, megestrol, or aminoglutethimide; and at least 2 weeks since prior bicalutamide or nilutamide
5. Radiation therapy and/or therapy with samarium must have been completed 4 weeks prior to first dose of therapy. Strontium therapy must have been completed at least 12 weeks prior to the first dose of therapy. The patient must have recovered from all treatment-related toxicities.
6. ECOG performance status ≤ 2
7. Able to swallow and retain oral medication

Exclusion Criteria:

1. Received prior chemotherapy (including estramustine phosphate [Estracyt]) for HRPC. Adjuvant chemotherapy (including docetaxel) is allowed provided that progression of disease occurred ≥ 6 months after the completion of adjuvant therapy.
2. Patients must not be receiving concurrent anti-androgen hormonal therapy for HRPC (LHRH directed therapies are acceptable to maintain castrate levels of testosterone).
3. Treatment with monoclonal antibody (e.g., VEGF targeting antibody) or prostate cancer vaccine within 45 days prior to the first dose of study treatment. Acute toxicities from prior therapy must have resolved to Grade ≤ 1.
4. Known history of or clinical evidence of central nervous system (CNS) metastases or leptomeningeal carcinomatosis
5. Active secondary malignancy or history of other malignancy within the last 5 years
6. Prior history of radiation therapy to ≥ 30% of the bone marrow
7. Peripheral neuropathy of ≥ Grade 2
8. Patients with malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel are excluded. Subjects with ulcerative colitis, inflammatory bowel disease, or partial or complete small bowel obstruction are also excluded.
9. Class 3 or 4 cardiac disease as defined by the New York Heart Association Functional Classification
10. Known active symptomatic fungal, bacterial and/or viral infection including active HIV. Note: screening for viruses is not required.
11. Psychiatric illness/social situations that would limit compliance with the study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2007-10; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
To evaluate and compare the two treatment arms with respect to overall survival (OS) | 33 months

SECONDARY OUTCOMES:
To evaluate and compare progression-free survival (PFS) in men with chemotherapy-naïve metastatic HRPC treated with AT-101 in combination with docetaxel and prednisone versus docetaxel and prednisone plus placebo. | 33 months
To determine the toxicities associated with oral AT-101 administered in combination with docetaxel and prednisone. | 28 months
To evaluate PSA and objective tumor response rate. | 28 months

CONTACTS AND LOCATIONS:
Overall Officials: Lance Leopold, MD, Study Director — Ascenta Therapeutics
Locations (35):
- United States (24):
  - Colorado Springs, Colorado
  - New Port Richey, Florida
  - Ocoee, Florida
  - Fishers, Indiana
  - Burnsville, Minnesota
  - Las Vegas, Nevada
  - Albuquerque, New Mexico
  - Las Cruces, New Mexico
  - Raleigh, North Carolina
  - Kettering, Ohio
  - Eugene, Oregon
  - Spartanburg, South Carolina
  - Amarillo, Texas
  - Arlington, Texas
  - Austin, Texas
  - Dallas, Texas
  - Denton, Texas
  - Midland, Texas
  - Paris, Texas
  - Webster, Texas
  - Fairfax, Virginia
  - Norfolk, Virginia
  - Kennewick, Washington
  - Vancouver, Washington
- Russia (11):
  - Barnaul
  - Engel's
  - Kazan'
  - Kursk
  - Kuzmolovsky
  - Moscow
  - Saint Petersburg
  - Sochi
  - Stavropol
  - Voronezh
  - Yekaterinburg

REFERENCES:
- [Derived] O'Neill AJ, Prencipe M, Dowling C, Fan Y, Mulrane L, Gallagher WM, O'Connor D, O'Connor R, Devery A, Corcoran C, Rani S, O'Driscoll L, Fitzpatrick JM, Watson RW. Characterisation and manipulation of docetaxel resistant prostate cancer cell lines. Mol Cancer. 2011 Oct 7;10:126. doi: 10.1186/1476-4598-10-126. PMID 21982118